CLINICAL TRIAL: NCT07179744
Title: A Multicenter, Prospective, Observational Study of Regional Radiotherapy Omission in Node Positive Patients With RecurIndex Low-risk Breast Cancer
Brief Title: Regional Radiotherapy Omission in Low-Risk Node Positive Breast Cancer
Status: Recruiting | Type: Observational
Sponsor: Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University (Other)
Collaborators: Sun Yat-sen University (Other)
Responsible Party: Sponsor
Other Study IDs: REOM
Record Dates: First submitted 2022-09-13; First posted 2025-09-18 (Actual); Last update posted 2025-09-18 (Actual); Status verified 2025-09

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Node Positive Breast Carcinoma: Omission of Regional Radiotherapy

SUMMARY:
The purpose of this study is to determine whether certain patients can safely omit regional lymph node radiotherapy. These women must have hormone-sensitive, Her2-negative tumors, have 1-3 positive axillary nodes and have RecurIndex low-risk.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years old, ≤ 70 years old.
* Eastern Cooperative Oncology Group (ECOG) ≤ 2.
* Postoperative pathology is clearly diagnosed as invasive breast cancer. Meet the clinical definition of low risk: ①Axillary lymph node micrometastasis (N1mic) or ②N1 patients who meet the following conditions at the same time,

  a）Age ≥ 40 years old, b）Vascular tumor thrombus (LVI) negative or allow few positive LVI (excluding extensive or massive LVI), c）ER positive (ER ≥ 1%) and HER2 negative (HER2 expression negative or + by IHC, or 2+ but negative by FISH).
* Postoperative pathological diagnosis of axillary lymph node status is any of the following: a. Sentinel lymph node biopsy or axillary lymph node dissection for micrometastasis (N1mic), b. Sentinel lymph node biopsy for 1-2 lymph node macrometastasis (N1sln), c. Sentinel lymph node biopsy + axillary lymph node dissection or simple axillary lymph node dissection for 1-3 lymph node metastasis (N1).
* The patient must have sufficient primary fresh frozen specimens or post- paraffin tissue sections for RecurIndex testing.
* Patients must have RecurIndex low risk obtained from testing of breast tumor tissue from a core biopsy or from the surgical specimen.
* The primary tumor and breast undergo breast-conserving surgery or total resection ± breast reconstruction (autologous/prosthetic).
* There must be adequate systemic examination (such as chest X-ray, B- ultrasound, CT, etc.) within 3 months before randomization of radiotherapy to confirm that there is no distant metastasis.
* Preoperative or radiotherapy should be performed within 12 months of randomization and must have mammography and/or MRI to confirm that there is no contralateral breast cancer.
* At least 4 courses of adjuvant chemotherapy with anthracycline or taxane should be completed after surgery.
* Radiotherapy must be performed sequentially after the completion of adjuvant chemotherapy, starting no later than 8 weeks after the end of chemotherapy.
* No previous history of malignant tumors, except for basal cell carcinoma of the skin.
* Signed an informed consent form.

Exclusion Criteria:

* Postoperative radiotherapy was confirmed as T3-4, N0, N2-3, M1 lesion staging before enrollment.
* Receive any new adjuvant therapy before surgery, including chemotherapy, endocrine therapy, targeted therapy or radiation therapy.
* Patients who underwent total mastectomy and only sentinel lymph node biopsy.
* Have a history of contralateral breast cancer.
* History of chest radiotherapy.
* combined with severe heart, lung, liver, kidney, hematopoietic, neurological diseases, and mental illness.
* History of autoimmune diseases such as scleroderma or active lupus erythematosus.
* pregnant and lactating patients.

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: pT1-2N1M0 breast cancer
Sampling Method: Probability Sample
Enrollment: 635 (Estimated)
Dates: Start 2022-07-06 (Actual); Primary Completion 2027-07-06 (Estimated); Study Completion 2032-07-05 (Estimated)

PRIMARY OUTCOMES:
Local-regional recurrence rate | 5 years
  defined as time between randomization and the time of any recurrence of ipsilateral chest, breast, regional lymph node recurrence, distant metastases, or death occurred

SECONDARY OUTCOMES:
Any first recurrence (AFR) | 5 years
  defined as any recurrence of ipsilateral chest, breast, regional lymph node recurrence, or distant metastases by Imaging or pathology
Local-regional recurrence free survival (LRFS) | 5 years
  defined as time between randomization and the time of any recurrence of ipsilateral chest, breast, regional lymph node recurrence, distant metastases, or death occurred
Recurrence free survival (RFS) | 5 years
  defined as time between randomization and the time of any recurrence of ipsilateral chest, breast, regional lymph node recurrence, distant metastases, or death occurred
Disease free survival (DFS) | 5 years
  defined as time between randomization and the time of disease recur or death occur
Beast cancer specific mortality (BCSM) | 5 years
  defined as time between randomization and the time of death occur specific due to breast cancer
Overall Survival (OS) | 5 years
  defined as time between randomization and the time of death occurred
Patient life quality measurement | 5 years
  At the screening period and after the end of radiotherapy, each group of patients was enrolled in the European Organisation for Research and Treatment of Cancer (EORTC) Quality of Life Questionnaire (QLQ) Cancer-30 (C30)
Patient life quality measurement | 5 years
  At the screening period and after the end of radiotherapy, each group of patients was enrolled in the European Organisation for Research and Treatment of Cancer (EORTC) Quality of Life Questionnaire (QLQ) Breast-23 (BR23)

CONTACTS AND LOCATIONS:
Locations (1):
- Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No